CLINICAL TRIAL: NCT01288066
Title: A Randomized Multicenter Study Comparing the Effectiveness of Hemi Versus Total Shoulder Arthroplasty in Patients With a Degenerative Joint Disease
Brief Title: Effectiveness of Hemi- Versus Total Shoulder Arthroplasty Using Implants of the "Epoca" System
Acronym: Epoca H vs T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AO Innovation Translation Center (Other)
Collaborators: Synthes GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Epoca Hemi vs. Total 2011
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
Keywords: Shoulder; Total arthroplasty; Hemiarthroplasty; Resurfacing; Glenoid; Constant score
MeSH Terms: conditions — Osteoarthritis | interventions — Hemiarthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemiarthroplasty (Other): Patients are treated with hemi shoulder arthroplasty with CE marked medical devices of the Epoca system.
  Interventions: Procedure: Hemiarthroplasty
- Total arthroplasty (Other): Patients are treated with total shoulder arthroplasty with CE marked medical devices of the Epoca system.
  Interventions: Procedure: Total arthroplasty

INTERVENTIONS:
Procedure: Hemiarthroplasty — Patients are treated with hemi shoulder arthroplasty with CE marked medical devices of the Epoca system. This procedure is a standard treatment for patients with a degenerative shoulder disease.
  Arms: Hemiarthroplasty
Procedure: Total arthroplasty — Patients are treated with total shoulder arthroplasty with CE marked medical devices of the Epoca system. This procedure is a standard treatment for patients with a degenerative shoulder disease.
  Arms: Total arthroplasty

SUMMARY:
The clinical question on whether or not to replace the glenoid component in patients with a degenerative shoulder disease, has not been answered yet in a randomized study with enough statistical power. In this study, patients are randomly allocated to a treatment with a hemi- or total shoulder arthroplasty using implants of the Epoca system. The primary objective is the comparison of pain and function between the treatment groups after 5 years using the Constant score.

DETAILED DESCRIPTION:
Shoulder arthroplasty is accepted as the treatment of choice for improved function with minimum pain in well-selected patients. A persistent discussion remains as to whether replacement of the glenoid (ie, total arthroplasty) should be performed. Possible advantages of glenoid replacement include decreased pain compared to hemiarthroplasty with a metal-on-bone articulation, increased stability due to the conforming glenoid component, and lateralization of the joint center providing improved range of motion and abduction strength. Potential complications of glenoid replacement are implant loosening and loss of glenoid bone stock.

If a hemiarthroplasty is performed, glenoid replacement and related complications are avoided. In addition, hemiarthroplasty requires less surgical time and is less expensive than total shoulder arthroplasty.

To date, there is no evidence to answer the clinical question on whether or not to replace the glenoid component in patients with a degenerative shoulder disease. In this study, both the stemmed Epoca humeral component (Epoca Stem) and the Epoca Resurfacing Head (Epoca RH) are included. While the stemmed prosthesis was developed both for nonreconstructable fractures and omarthroses, the humeral resurfacing head implant was designed specifically for use in degenerative diseases of the shoulder joint.

This randomized multicenter study aims to compare the efficacy of hemi versus total shoulder arthroplasty using Epoca RH or Epoca Stem in patients with degenerative joint diseases. The primary aim of the present study is to demonstrate that the Constant score assessing shoulder function and pain is higher in the patient group treated with total arthroplasty compared to the hemiarthroplasty group after 5 years. The secondary aims of the study are to assess differences in the Shoulder Pain and Disability Index (SPADI), duration of surgery, rates of local and general adverse events and relationship to the device or treatment under investigation, survivorship of the implants, and quality of life after 6 months, 1, 3 and 5 years between the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Primary or secondary omarthrosis (eg, rheumatoid arthritis, avascular head necrosis)
* Glenoid morphologic type A1, A2 or B1 according to Walch
* Ability to understand the content of the patient information / informed consent form and to participate in the clinical investigation
* Written informed consent

Exclusion Criteria:

Preoperative:

* Posttraumatic omarthrosis
* Biconcave aspect of glenoid (Walch type B2)
* Retroversion of glenoid more than 25° (Walch type C)
* "Epoca Reko" prosthesis
* Humerus fractures
* Patients with a severe systemic disease: class III-IV according to the American Society of Anaesthesiologists physical status classification (ASA)
* Substance abuse that would preclude reliable assessment
* Pregnancy
* Prisoners
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Intraoperative:

* Full thickness tear of rotator cuff
* Indication for hemiarthroplasty only
* Indication for total arthroplasty only
* Intraoperative decision to use implants other than Epoca

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-09; Primary Completion 2024-06 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
The Constant score assessment of shoulder function and pain | Baseline to 5 years postsurgery
  The primary outcome measure is the difference between the Constant score assessment of shoulder function and pain at baseline and 5 years after surgery. This difference is assessed for each individual patient.

SECONDARY OUTCOMES:
Constant score | 6 months, 1 year, 3 years
Shoulder Pain and Disability Index (SPADI) | 6 months, 1 year, 3 years, 5 years
Duration of surgery | 1-2 days
Numbers of adverse events | Baseline to 5 years follow-up
Survivorship of implants | Baseline to 5 years follow-up
Quality of life related to health | Baseline, 6 months, 1 year, 3 years, 5 years
  Quality of life is assessed using the Euroqol - 5 Dimensions (EQ-5D) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Suedkamp, MD, Principal Investigator — Universitätsklinikum Freiburg, Deutschland
Locations (4):
- Medizinische Universität, Innsbruck, Austria
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Region Hannover GmbH, Klinikum Agnes-Karll Laatzen, Laatzen
- Universitetssjukhuset Ortopedicentrum i Östergötland, Linköping, Sweden